CLINICAL TRIAL: NCT01828281
Title: A Randomized Controlled Study on the Effects of Continuous Positive Airway Pressure (CPAP) on Visceral Fat Thickness, Carotid Intima-media Thickness and Adipokines in Patients With Obstructive Sleep Apnoea Syndrome (OSAS)
Brief Title: Effects of CPAP on Visceral Fat Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VF-CPAP
Record Dates: First submitted 2013-04-08; First posted 2013-04-10 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic CPAP (Active Comparator): Therapeutic CPAP
  Interventions: Device: CPAP
- control (Sham Comparator): subtherapeutic CPAP using 4 cm water
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — All subjects will undergo ultrasound examination of the abdomen the day after overnight polysomnography (PSG) and then at 3 months after completion of therapeutic or subtherapeutic CPAP treatment of 4 cm water.

SUMMARY:
We hypothesize that patients with untreated OSAS will have more visceral fat, fatty liver and increased carotid artery thickness whereas treatment with CPAP may reduce the mesenteric and liver fat, plasma lipids, carotid artery thickness.

DETAILED DESCRIPTION:
This proposed randomized control trial (RCT) will compare the effects of therapeutic CPAP versus subtherapeutic CPAP in patients newly diagnosed with OSA with reference to visceral fat especially mesenteric fat thickness, liver fat, carotid artery intima media thickness (IMT), lateral pharyngeal wall (LPW) thickness, plasma lipids and adipokines over a treatment period of 3 months. The results of this study will advance our understanding of the relative role of OSA and obesity in the pathogenesis of metabolic syndrome (MetS) and whether CPAP therapy can improve these metabolic dysregulation.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients with OSA of apnea hypopnea index (AHI) >= 5/hr

Exclusion Criteria:

* Recent or past history of myocardial infarction/stroke/heart failure, unstable angina, underlying malignancy,
* patients with clinical features of any active infection
* those who require urgent CPAP treatment because of associated respiratory failure or to prevent job loss through excessive daytime sleepiness (eg professional drivers, those handling dangerous machinery)
* moderate to severe valvular heart disease, cardiomyopathy, and previous diagnosis of OSA and/or previous use of CPAP therapy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui David, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Respiratory Division, Hong Kong, China

REFERENCES:
- [Derived] Ng SS, Liu EK, Ma RC, Chan TO, To KW, Chan KK, Ngai J, Yip WH, Ko FW, Wong CK, Hui DS. Effects of CPAP therapy on visceral fat thickness, carotid intima-media thickness and adipokines in patients with obstructive sleep apnoea. Respirology. 2017 May;22(4):786-792. doi: 10.1111/resp.12963. Epub 2016 Dec 9. PMID 27933703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients referred by general practitioners to the respiratory clinics with clinical suspicion of sleep-disordered breathing over the period 17 Feb 2012 to 30 Oct 2013. Overnight polysomnography (PSG) were performed as inpatient at the hospital.
Pre-assignment Details: 51 subjects were excluded as 26 had AHI <5 events/hour and 25 were not interested in continuing study.
Groups:
- Therapeutic CPAP: The continuous positive airway pressure (CPAP) level for each patient in the arm was set at the minimum pressure needed to abolish snoring, obstructive respiratory events and airflow limitation for 95% of the night, as determined by the overnight CPAP titration study.
Period: Overall Study
Arm/Group | Therapeutic CPAP | Control
Started | 45 | 45
Completed | 44 | 45
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Therapeutic CPAP: The CPAP level for each patient in the arm was set at the minimum pressure needed to abolish snoring, obstructive respiratory events and airflow limitation for 95% of the night, as determined by the overnight CPAP titration study.
- Total: Total of all reporting groups
Arm/Group | Therapeutic CPAP | Control | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (10.1) | 48.7 (9.0) | 49.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 32 | 31 | 63
Neck circumference (cm) [Mean (Standard Deviation); unit: cm] | 40.7 (11.3) | 39.1 (3.7) | 39.9 (7.5)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 28.2 (3.9) | 28.2 (4.5) | 28.2 (4.1)
Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — minimum score of the scale is 0 and maximum is 24. The higher the score the sleepier the subject is.
  units on a scale | 12.4 (5.9) | 11.3 (4.7) | 11.9 (5.1)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 132.1 (16.4) | 129.4 (21.6) | 130.2 (18.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 83.8 (12.9) | 83.9 (14.1) | 83.8 (13.6)
Apnea hypopnea index (AHI) (event/hour) [Mean (Standard Deviation); unit: event/hour] | 30.6 (21.4) | 35.2 (25.5) | 33.2 (22.4)
Mesenteric fat thickness [Mean (Standard Deviation); unit: cm] | 0.97 (0.28) | 0.98 (0.26) | 0.98 (0.27)
Adiponectin [Mean (Standard Deviation); unit: ug/ml] | 25.2 (25.9) | 22.5 (23.8) | 24.1 (23.9)

OUTCOME MEASURES:

1. Primary Outcome: Mesenteric Fat Thickness
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Control: subtherapeutic CPAP using 4 cm water
  CPAP: All subjects will undergo ultrasound examination of the abdomen the day after overnight PSG and then at 3 months after completion of therapeutic or subtherapeutic CPAP treatment of 4 cm water.
Arm/Group | Therapeutic CPAP | Control
Number analyzed (Participants) | 45 | 45
cm | 0.96 (0.16) | 0.94 (0.13)

2. Secondary Outcome: Mean Changes in Adiponectin Over 3 Months
Description: Mean changes in Adiponectin from baseline to 3 months.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Therapeutic CPAP | Control
Number analyzed (Participants) | 45 | 45
ug/ml | 23.63 (23.44) | 29.78 (38.07)

3. Other Pre Specified Outcome: Mean Hours of CPAP Usage Per Day
Description: Mean Hours of CPAP usage per day in those who continue to use CPAP during the three month period.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Therapeutic CPAP | Control
Number analyzed (Participants) | 45 | 45
hours | 4.18 (2.07) | 4.11 (1.99)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Therapeutic CPAP: The CPAP level for each patient in the therapeutic CPAP arm was set at the minimum pressure needed to abolish snoring, obstructive respiratory events and airflow limitation for 95% of the night, as determined by the overnight CPAP titration study.
Arm/Group | Therapeutic CPAP | Control
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No